CLINICAL TRIAL: NCT04561700
Title: Nutritive Sucking Patterns in Premature Infants: A Randomized Trial
Brief Title: Nutritive Sucking Patterns in Premature Infants
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unfunded
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Ariel A. Salas, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 300004412
Record Dates: First submitted 2020-09-05; First posted 2020-09-24 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Premature; Light-For-Dates Without Mention of Fetal Malnutrition, Unspecified; Feeding Patterns
MeSH Terms: conditions — Premature Birth; Feeding Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reporting of sucking patterns captured by Instrumented Bottle (Experimental): Weekly reporting on objective measurements of sucking activity during oral feeding
  Interventions: Diagnostic Test: Reporting of sucking patterns captured by Instrumented Bottle
- Control (Sham Comparator): Weekly reporting on traditional measurements of sucking activity during oral feeding (no objective measurements reported)
  Interventions: Diagnostic Test: Control

INTERVENTIONS:
Diagnostic Test: Reporting of sucking patterns captured by Instrumented Bottle — In the intervention group, data on nutritive sucking and feeding cues captured by the Instrumented Bottle will be made available to speech therapists to document the feeding session and provide written recommendations in their weekly report.
  Arms: Reporting of sucking patterns captured by Instrumented Bottle
Diagnostic Test: Control — In the control group, the information captured by the Instrumented Bottle will not be made available to speech therapists and therefore, will not be used to document a feeding session or provide weekly recommendations.
  Arms: Control

SUMMARY:
In this pilot trial, the investigators will determine the feasibility of monitoring nutritive sucking patterns to facilitate the transition from tube to oral feeding in extremely-low-birth weight (ELBW) infants

DETAILED DESCRIPTION:
In this parallel-group randomized controlled trial, ELBW infants (birthweight < 1000 grams) will be randomly assigned in a 1:1 ratio to either weekly reporting on objective measurements of sucking activity during oral feeding (intervention group) or usual care without information on sucking activity (control group).

ELIGIBILITY:
Inclusion Criteria:

* Birthweight < 1000 grams
* Gestational age < 32 weeks of gestation
* Full enteral feeding established before or on postnatal day 21
* Oral feeding initiated before or at 33 weeks of postmenstrual age

Exclusion Criteria:

* Major congenital/chromosomal anomalies
* Patent ductus arteriosus causing significant cardiovascular symptoms
* History of necrotizing enterocolitis stage 2 or greater

Ages: 7 Days to 60 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Time to independent oral feeding | Birth to 120 days
  Time interval in days from introduction of oral feeding to full independent oral feeding

SECONDARY OUTCOMES:
Postnatal age at discharge | Birth to 120 days
  Age in days at the time of hospital discharge
Length of hospital stay | Birth to 120 days
  Total number of hospitalization days
Growth rate during the transition from tube to oral feeding | Birth to 120 days
  Weekly weight gain in g/kg/day
Tube feeding events per day during the transition from tube to oral feeding. | Birth to 120 days
  Daily count of tube feeding events

CONTACTS AND LOCATIONS:
Overall Officials: Ariel A. Salas, MD, MSPH, Principal Investigator — University of Alabama at Birmingham